CLINICAL TRIAL: NCT04226183
Title: Natural Antioxidant Intake After Exercise Can Reduce Malondialdehyde (MDA) Level in the Third Trimester of Pragnancy
Brief Title: Natural Antioxidant Intake After Exercise Can Oxidative Stress in the Third Trimester of Pragnancy
Acronym: MDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Indonesia-MoH (Other Government)
Responsible Party: Principal Investigator, Dr. Ocktariyana, SST, M.Kes, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: qwery123
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Stress Oxidative
Keywords: Antioxidants; Malondialdehyde level; the third trimester of pregnancy; exercise; anti oxidant; stress oxidative
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: There were 24 prenatal pregnant women and separated to 3 groups, which were 8 prenatal pregnant women without exercise as a control group, 8 prenatal pregnant women with exercise as a positive control group and 8 prenatal pregnant women with exercise and consume natural antioxidants after exercise as a treatment group. The antioxidant compounds given in this study were guava juice that contains vitamin C.
Who Masked: Care Provider, Investigator
Masking Description: care provider is a midwifery as a intructure of excercise and measure of each pregnant participans condition.
  investigator is controling all reseach procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (No Intervention): pregnant women without pregnancy workout and consume guava juice
- positive control group (Experimental): prenatal pregnant women with pregnancy workout but not consume guava juice
  Interventions: Other: pregnancy workout
- treatment group (Experimental): prenatal pregnant women with pregnancy workout and consume guava juice
  Interventions: Other: pregnancy workout

INTERVENTIONS:
Other: pregnancy workout — Procedure of pregnancy workout has been legalized by the Ministry of Health of Indonesia act 2014 No.97.
  100 ml fresh guava juice without sugar
  Other Names: fresh Guava juice
  Arms: positive control group; treatment group

SUMMARY:
Pregnancy is a condition that increased requirements of energy and oxygen, and if this condition is not maximally that can lead oxidative stress and produce free radicals which is affect in the pregnancy process. Malondialdehyde (MDA) level in pregnant women is higher than non-pregnant women. Exercise is one way to neutralize the free radical. The aim of this study was analyzed effect of treatment natural antioxidants after exercise which was pregnancy workout to MDA level in the third trimester of pregnancy.

This study was a true experimental study. There were 24 prenatal pregnant women and separated to 3 groups, which were 8 prenatal pregnant women without pregnancy workout as a control group, 8 prenatal pregnant women with pregnancy workout but without natural antioxidant consume as a positive control group, and 8 prenatal pregnant women with natural antioxidant consume after pregnancy workout as a treatment group. The antioxidant compounds given in this study were guava juice that contains vitamin C. MDA levels was analyzed by spectrophotometric. Comparison between groups was done by one way ANOVA test.

DETAILED DESCRIPTION:
Pregnancy is a condition that is vulnerable to all kinds - stress resulting in changes in physiology and metabolic function. In pregnancy there is also an increase in energy and oxygen requirements.

The metabolic process can increase require of the oxygen and if it is not available as well as unmaximal used can causes the formation of oxidative stress and produces excessive free radicals which ultimately, that affected in the saferity of a pregnancy process. The imbalance between antioxidants and free radicals in pregnancy prosses are causes pathological and complications changes in pregnancy. This kind of biochemical marker of antioxidants and oxidants is very useful in observing complications that may arise in pregnancy.

Treatment given is expected to eliminate complaints that arise while exercise during pregnancy can prevent the formation of free radicals, but exercise must be given in accordance with the ability of pregnant women.

Physical exercise or exercise in pregnancy can maintain excess weight gain, prevent diabetes, hypertension, and shorten labor time. Sports is one way to neutralize the formation of free radicals because by doing physical activity, excessive oxygen can be used to produce energy.

Increased free radicals are characterised by an increase of malondialdehyde (MDA) as a biochemical markers. Malondialdehyde (MDA) which is the output of lipid peroxidation prosses that measured to determine the presence of oxidative stress due to damage by free radicals. The resent study was found that MDA levels in pregnant women were higher compared to non-pregnant women. Increased MDA levels are in line with the increase in gestational age, from the first, second, and third trimesters. Study was also found that there was a significant increase in MDA levels accompanied by a decrease in non-enzymatic antioxidants, such as Vitamin-E, Vitamin-C, and Vitamin-A in pregnant women with hypertension. Moreover this study assums that was "Giving Antioxidant to decrease Malondialdehyde (MDA) in the third trimester of pregnancy". futher more the aims of this study was analyzed effect of natural antioxidants treatment after exercise to MDA level in the third trimester of pregnancy.

This study was a experimental study. This study was located in the several clinics midwife practice, Community Health Centers (Puskesmas) in Palembang and Bio Sains Riset Laboratory Palembang from August to October 2016.

the study was approved informed consent from all participans as well as ethical clearance approval number is 007/UP-ETIK/I/2016. This study was obtained 24 prenatal pregnant women that separated to 3 groups, which were 8 prenatal pregnant women without pregnancy workout exercise as a control group, 8 prenatal pregnant women with pregnancy workout exercise as a positive control group and 8 prenatal pregnant women with consume natural antioxidants after pregnancy workout exercise as a treatment group.

The antioxidant compounds given in this study were natural vitamin C from 100 ml guava juice without additionaly sugar, 5 cc syringe, cotton, alcohol, syringe, hanscoon, EDTA tube, serum, TCA 5%, Na thiobarbiturat 0,65%, MDA standart, and aquades.

Spectrophotometric assay used to measure the MDA levels in the Bio Sains Riset Laboratory, Palembang and followed the essay of protocol kit from manufacture.

Comparison between groups used by one way ANOVA test, that was considered significant if p < 0.05. All statistical analyses were done by SPPS for Windows version 16.0.

ELIGIBILITY:
Inclusion Criteria:

* Approve as a subject of review and sign in an informed consent
* Approve to take 3 ml of whole blood.
* Ages 20-30 years
* Hemoglobin levels higher than 11 gr%
* Third trimester of pregnancy
* Healthy condition during reseach

Exclusion Criteria:

* Anemia
* Pathologies condition during pregnant
* Allergic
* Disability

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-02-03 (Actual); Primary Completion 2016-08-26 (Actual); Study Completion 2016-10-17 (Actual)

PRIMARY OUTCOMES:
MDA level | 7 days.
  Malondialdehyde (MDA) levels is stress oxidative marker. MDA level messured with spectrophotometric assay. at Bio Sains Riset Laboratory, Palembang. Firstly, Mix 0.5ml blank + 0.5 ml standard and 0.5 ml serum using vortex mixer. Centrifuge for 10 minutes, with a speed of 2000 rpm, and Pipette 1 ml each filtrate and after that put it in boiling water bath for 30 minutes, then chill and read the absorbance with a spectrophotometer with a wavelength of 550 nm.

CONTACTS AND LOCATIONS:
Overall Officials: Ocktariyana Ocktariyana, Principal Investigator — Ministry of health, Health Polytechnic, Palembang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nazari A, Dirandeh E, Ansari-Pirsaraei Z, Deldar H. Antioxidant levels, copper and zinc concentrations were associated with postpartum luteal activity, pregnancy loss and pregnancy status in Holstein dairy cows. Theriogenology. 2019 Jul 15;133:97-103. doi: 10.1016/j.theriogenology.2019.04.034. Epub 2019 Apr 30. PMID 31078069
- [Result] Patil SB, Kodliwadmath MV, Kodliwadmath SM. Correlation between lipid peroxidation and non-enzymatic antioxidants in pregnancy induced hypertension. Indian J Clin Biochem. 2008 Jan;23(1):45-8. doi: 10.1007/s12291-008-0011-9. Epub 2008 Mar 6. PMID 23105719